CLINICAL TRIAL: NCT03844048
Title: An Extension Study of Venetoclax for Subjects Who Have Completed a Prior Venetoclax Clinical Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19-388; 2022-501522-38-00 (Other: EU CT)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia; Acute Myeloid Leukemia; Multiple Myeloma; Non-Hodgkin's Lymphoma; Acute Lymphoblastic Leukemia; Cancer
Keywords: Chronic Lymphocytic Leukemia (CLL); Acute Myeloid Leukemia (AML); Multiple Myeloma (MM); Non-Hodgkin's Lymphoma (NHL); Acute Lymphoblastic Leukemia (ALL); Cancer; Venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Multiple Myeloma; Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Venetoclax (Experimental): Venetoclax at the same dose administered to each subject during the previous study in which they were enrolled.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — oral; film-coated tablets or tablets for oral suspension
  Other Names: ABT-199; Venclexta

SUMMARY:
The purpose of this extension study is to provide venetoclax and obtain long-term safety data for subjects who continue to tolerate and derive benefit from receiving venetoclax in ongoing studies.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been enrolled and dosed in an ongoing venetoclax study and continues to tolerate and derive benefit from the study drug.
* Male subject agrees to refrain from sperm donation.
* Female subjects must not be pregnant or breastfeeding.

Exclusion Criteria:

- None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | From first dose of study drug until 30 days following last dose of study drug (up to approximately 5 years).
  An adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (56):
- United States (7):
  - University of Arizona Cancer Center - Tucson /ID# 210548, Tucson, Arizona
  - UCLA Santa Monica Hematology Oncology /ID# 210551, Los Angeles, California
  - Ingalls Memorial Hosp /ID# 210553, Harvey, Illinois
  - Dana-Farber Cancer Institute /ID# 215360, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 231132, Ann Arbor, Michigan
  - Dartmouth-Hitchcock Medical Center /ID# 210555, Lebanon, New Hampshire
  - Swedish Cancer Institute /ID# 213120, Seattle, Washington
- Australia (6):
  - Royal Prince Alfred Hospital /ID# 239557, Camperdown, New South Wales
  - St George Hospital /ID# 225589, Kogarah, New South Wales
  - Liverpool Hospital /ID# 225591, Liverpool, New South Wales
  - Peter MacCallum Cancer Ctr /ID# 210559, Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 239480, Murdoch, Western Australia
  - Perth Blood Institute Ltd /ID# 225592, Nedlands, Western Australia
- Duplicate_Medizinische Universitaet Graz /ID# 223817, Graz, Styria, Austria
- Cliniques Universitaires UCL Saint-Luc /ID# 224327, Brussels, Brussels Capital, Belgium
- CHUQ- Hôpital de l'Enfant-Jesus /ID# 224616, Québec, Quebec, Canada
- Denmark (2):
  - Rigshospitalet /ID# 224213, Copenhagen Ø, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 224214, Aarhus, Central Jutland
- France (2):
  - CHU Grenoble - Hopital Michallon /ID# 240497, La Tronche, Isere
  - HCL - Hopital Lyon Sud /ID# 213508, Pierre-Bénite, Rhone
- Greece (2):
  - General Hospital of Athens Laiko /ID# 224087, Athens, Attica
  - General Hospital of Thessaloniki George Papanikolaou /ID# 224088, Thessaloniki
- Queen Mary Hospital /ID# 224944, Hong Kong, Hong Kong
- Beaumont Hospital /ID# 225165, Dublin, Ireland
- Japan (4):
  - Kobe City Medical Center General Hospital /ID# 241518, Kobe, Hyōgo
  - Duplicate_National Hospital Organization Mito Medical Center /ID# 241986, Higashi Ibaraki-gun, Ibaraki
  - Okayama Medical Center /ID# 241517, Okayama, Okayama-ken
  - National Cancer Center Hospital /ID# 241516, Chuo-ku, Tokyo
- Mexico (2):
  - Centro de Investigacion Clínica Chapultepec SA de CV /ID# 227018, Morelia, Michoacán
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 227017, Monterrey, Nuevo León
- New Zealand (3):
  - Aotearoa Clinical Trials /ID# 225596, Papatoetoe, Auckland
  - North Shore Hospital /ID# 225597, Takapuna, Auckland
  - Wellington Regional Hospital /ID# 225593, Newtown, Wellington Region
- Poland (3):
  - Duplicate_Pratia MCM Krakow /ID# 218561, Krakow, Lesser Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii /ID# 225478, Warsaw, Masovian Voivodeship
  - SP ZOZ Zespol Szpitali Miejskich w Chorzowie /ID# 225474, Chorzów, Silesian Voivodeship
- IPO Lisboa FG, EPE /ID# 225072, Lisbon, Portugal
- Russia (2):
  - Federal State Budgetary Scientific Institution N.N. Blokhin /ID# 225194, Moscow, Moscow
  - Regional Oncological Dispensary /ID# 225195, Penza, Penza Oblast
- Samsung Medical Center /ID# 240882, Seoul, Seoul Teugbyeolsi, South Korea
- Hospital Universitario Fundacion Jimenez Diaz /ID# 225476, Madrid, Spain
- Duplicate_Skane University Hospital Lund /ID# 224747, Lund, Skåne County, Sweden
- Taiwan (2):
  - National Taiwan University Hospital /ID# 224946, Taipei City, Taipei
  - China Medical University Hospital /ID# 224945, Taichung
- Turkey (Türkiye) (3):
  - Ankara Univ Medical Faculty /ID# 225043, Ankara
  - Istanbul University Istanbul Medical Faculty /ID# 225045, Istanbul
  - Vehbi Koc vakfi Amerikan Hasta /ID# 225046, Istanbul
- Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council /ID# 240575, Dnipro, Ukraine
- United Kingdom (8):
  - Derriford Hospital and the Royal Eye Infirmary /ID# 218731, Plymouth, Devon
  - Leicester Royal Infirmary /ID# 240468, Leicester, England
  - University College London Hospital /ID# 240467, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 225161, Southampton, Hampshire
  - Blackpool Teaching Hospitals NHS Foundation Trust /ID# 225163, Blackpool
  - Clatterbridge Cancer Centre - Liverpool /ID# 218736, Liverpool
  - King's College Hospital NHS Foundation Trust /ID# 218735, London
  - The Royal Wolverhampton NHS Trust /ID# 225164, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-388